CLINICAL TRIAL: NCT07229742
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Study to Evaluate the Efficacy and Safety of SHR-2173 Injection in Patients With Active Lupus Nephritis
Brief Title: A Phase II Clinical Study on the Efficacy and Safety of SHR-2173 Injection in the Treatment of Patients With Active Lupus Nephritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-2173-204
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Active Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-2173 Injection Group (Experimental)
  Interventions: Drug: SHR-2173 Injection
- SHR-2173 Injection Placebo Group (Placebo Comparator)
  Interventions: Drug: SHR-2173 Injection Blank Preparation

INTERVENTIONS:
Drug: SHR-2173 Injection — SHR-2173 injection.
  Arms: SHR-2173 Injection Group
Drug: SHR-2173 Injection Blank Preparation — SHR-2173 injection blank preparation.
  Arms: SHR-2173 Injection Placebo Group

SUMMARY:
The study is a Phase II clinical trial to evaluate the efficacy and safety of SHR-2173 in patients with lupus nephritis (LN). It adopts a randomized, double-blind, placebo-controlled, multicenter trial design.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years (inclusive) at informed consent signing, regardless of sex;
2. Body weight ≥ 40.0 kg and body mass index (BMI) ≥ 16 kg/m² to ≤ 28 kg/m² at screening;
3. Diagnosed with systemic lupus erythematosus (SLE) per 1997 ACR criteria or 2019 EULAR/ACR classification criteria;
4. Positive antinuclear antibody (titer ≥ 1:80) and/or anti-dsDNA antibody and/or anti-Sm antibody at screening;
5. Histologically confirmed active lupus nephritis (LN) class III or IV ± class V by renal biopsy, per 2018 International Society of Nephrology/Renal Pathology Society (ISN/RPS) standards within 1 year preceding or during screening.

Exclusion Criteria:

1. Received renal dialysis within 12 months preceding screening, or anticipated requirement for dialysis/renal transplantation within 6 months post-enrollment;
2. Renal biopsy demonstrating > 50% globally sclerosed glomeruli;
3. Active severe/unstable neuropsychiatric SLE (NPSLE);
4. Catastrophic antiphospholipid syndrome (APS) within 12 months pre-screening, or APS-related thrombotic events (except non-catastrophic/mild APS cases with stable anticoagulation ≥12 weeks prior to screening);
5. Non-LN renal diseases potentially confounding disease assessment (e.g., diabetic nephropathy per investigator judgment);
6. Inflammatory/autoimmune diseases beyond SLE/LN that may interfere with efficacy/safety interpretation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
The ratio of 24-hour urine protein-creatinine ratio (24-hour UPCR) to the baseline. | At Week 24.

SECONDARY OUTCOMES:
The proportion of subjects achieving complete renal response (CRR). | At Week 24 and Week 52.
The proportion of subjects achieving partial renal response (PRR). | At Week 24 and Week 52.
The proportion of subjects achieving at least 50% improvement in 24-hour UPCR compared to the baseline. | At Week 24 and Week 52.
The proportion of subjects achieving at least 25% improvement in 24-hour UPCR compared to the baseline. | At Week 24 and Week 52.
The proportion of subjects whose 24-hour UPCR was less than 0.5 g/g. | At Week 24 and Week 52.
The proportion of subjects whose 24-hour UPCR was less than 0.7 g/g. | At Week 24 and Week 52.
The proportion of subjects taking prednisone or the equivalent dose of glucocorticoids ≤ 5 mg/day. | At Week 24 and Week 52.
The proportion of subjects taking prednisone or the equivalent dose of glucocorticoids ≤ 7.5 mg/day. | At Week 24 and Week 52.
The changes in the Chronic Disease Treatment Function Assessment - Fatigue Scale (FACIT) score relative to the baseline. | At Week 24 and Week 52.
Adverse events (AEs). | Up to 52 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The General Hospital of the Eastern Theater Command of the People's Liberation Army of China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided